CLINICAL TRIAL: NCT05881655
Title: A Prospective Clinical Trial on Slow Myopia Progression With Two Different Irradiance Light at Baseline and Dynamic Changes at Follow-up
Brief Title: Slow Myopia Progression With Different Irradiance Light
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Airdoc Technology Co., Ltd. (Industry)
Collaborators: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Airdoc MPC
Record Dates: First submitted 2023-05-20; First posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Myopia, Progressive
MeSH Terms: conditions — Myopia, Degenerative | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Group 1 (Experimental): With 1.2mW lighting power of red light at wavelenth of 650nm and wearing H.A.L.T lens to control myopia.
  Interventions: Device: Airdoc Red Lighting Device; Device: Special Spectacles to Control Myopia
- Study Group 2 (Experimental): With 0.6mW lighting power of red light at wavelenth of 650nm and wearing H.A.L.T lens to control myopia.
  Interventions: Device: Airdoc Red Lighting Device; Device: Special Spectacles to Control Myopia
- Control Group (Placebo Comparator): Wearing H.A.L.T lens to control myopia only.
  Interventions: Device: Special Spectacles to Control Myopia

INTERVENTIONS:
Device: Airdoc Red Lighting Device — A medical device with ultra low lever laser irradiance of 0.6mW or 1.2mW at the surface of cornea. And the therapy lasts 3 minutes with the 4 hours or more interval of break.
  Other Names: Repeated Red Light, Low Lever Laser Therapy, Low Intensity Light Therapy, Photobiomodulation Therapy, Seconee, 650nm Red Light
  Arms: Study Group 1; Study Group 2
Device: Special Spectacles to Control Myopia — Customer designed power and fitting to each subject for all the study periods.
  Other Names: Essilor® Stellest™ Lenses; H.A.L.T lens

SUMMARY:
It is a prospective clinical control study on red light control myopia with specail design spectacles for 75 children in 3 groups. Study Groups with two different powers of 0.6 mW and 1.2 mW at wavelength of 650nm. The control group is to wear the same brand and design spectalces as those two study groups. In addition, the progression of myopia is usually accompanied by the changes in a variety of ocular parameters, such as refractive error, reduced submacular choroidal thickness, and prolonged length of the ocular axis length.The goal is to test which power (1.2mW and 0.6mW) is better in myopic children for 3 month's follow-up and also to test how to get better result with the increaing or decreasing lighting power for the total 6 month follow-up results .

DETAILED DESCRIPTION:
It is a prospective clinical control study on red light control myopia with specail design spectacles for 75 children in 3 groups. Each group has 25 myopic children. Study Groups with two different powers of 0.6 mW and 1.2 mW at wavelength of 650nm are randomized to be allocated into the 3 groups. The control group is to wear the same brand and design spectalces as those two study groups. In addition, the progression of myopia is usually accompanied by the changes in a variety of ocular parameters, such as refractive error, reduced submacular choroidal thickness, and prolonged length of the ocular axis length. All groups will be wearing a special lens named by Stellest with high aspherical lens design.

ELIGIBILITY:
Inclusion Criteria:

* 6~12 years old
* Refractive Error of Myopia within -0.50 D~-5.00 D, Anisometropia less or equal to 2.00D, The best corrected vision acuity is better or equal to 0.8 （decimal record).
* Written consent formed with supervisions and children with 6 month follow-up.

Exclusion Criteria:

* Photophobia or allergy to any cycloplegic eyedrops (such as tropcaine, cyclopentolate).
* Lesions in fundus or any part of eyeball with abnormal corrected vision such as keratoconus.
* Strabisumus with angles large or equal to 5 prism dioper.
* With other myopia control device such as atropine, Orthokeratology, Misight lens or other myopia control device.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change of Ocular Axial length elongation at follow-up from Baseline (mm) | 3-month
  Measured with IOLmaster 500 or Lenstar at follow-up from baseline
Mean Change of Ocular Axial length elongation at follow-up from Baseline (mm) | 6-month
  Measured with IOLmaster 500 or Lenstar at follow-up from baseline

SECONDARY OUTCOMES:
Mean Change of Refractive Error at follow-up from Baseline (mm) | 3-month
  Measured with autorefractor; Spherical Equivalence is calculated.
Mean Change of Refractive Error at follow-up from Baseline (mm) | 6-month
  Measured with autorefractor; Spherical Equivalence is calculated according to the formular of SE=Spherical +1/2 * Cyclinder Diopter.
Mean Change of Choroidal Thickness (um) | 3-month
  Measured with Optical Coherence Topography (OCT)
Mean Change of Choroidal Thickness (um) | 6-month
  Measured with Optical Coherence Topography (OCT)
Change of Fundus | 6-month
  Mesured with color fundus camera with Artificial Intelligence Database

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, MD, PHD, Principal Investigator — Shanghai Children's Medical Center
Locations (1):
- Shanghai Children Medical Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No